CLINICAL TRIAL: NCT01023165
Title: Multicenter Trial to Evaluate the Effects of Intensive Bolus Intravenous Insulin Delivery on Metabolic Integrity in Type 1 and Type 2 Diabetics Who Despite Tight Control and Proper Diet Still Suffer From Metabolic Problems
Brief Title: Effects of Intensive Bolus Intravenous Insulin Delivery on Metabolic Integrity in Type 1 and Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Global Infusion and Aspiration Systems, LLC (Other)
Responsible Party: Michael Cockrell MD, Global Infusion and Aspiration Systems, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI-001
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus; Metabolic Integrity
Keywords: Diabetes Mellitus; Metabolic Integrity; Intravenous Bolus Insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin, Regular, Human; Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV bolus insulin, metabolic integrity (Experimental): Diabetic patients will complete diagnostic testing and complete quality of life questionnaires at baseline and every six months thereafter while enrolled in the study to monitor and assess progress with metabolic integrity and complications resulting from their diabetes. Comparisons will be performed on lab values performed at baseline and every six months thereafter. Supervising physician may request testing be performed more frequently as deemed medically necessary, testing may include retinal photography, nerve conduction and labs. Meds and medical intervention information is collected weekly at the Intravenous Bolus Insulin treatment sessions. An annual evaluation is performed to review clinical data collected and evaluate progress for analysis and comparison.
  Interventions: Procedure: Humulin, Humalog, Novolog

INTERVENTIONS:
Procedure: Humulin, Humalog, Novolog — Supervising Physician reviews patient activation after intravenous bolus insulin treatment each week and adjusts the amounts of insulin and carbohydrates to be given in the next treatment session based on patient treatment outcomes.

SUMMARY:
The purpose of this study is to determine if restoring normal metabolic function in patients with type 1 or type 2 diabetes can improve the impact of the consequences of diabetic complications on the overall health and quality of life for diabetic patients.Patients are treated once per week with intensive bolus intravenous insulin delivery mimicking normal insulin secretions in a non diabetic individual. Baseline and periodic diagnostic tests are performed and questionnaires completed to evaluate and monitor progress and outcomes.

DETAILED DESCRIPTION:
It is known that the glucose metabolic pathway is the primary fuel generator to the brain, nerve tissue, heart, vascular tissue, eyes, kidneys and the liver. Deficient metabolism state as seen in the glucose metabolism experienced in many diabetic patients can lead to complications. These damaging effects are exacerbated by altered cellular metabolites, specifically the increase in catabolic and decrease in anabolic factors. It has been shown over the past 20 years that normalization of metabolism in diabetic patients can be accomplished by mimicking the normal endogenous insulin pattern from the pancreas. Intensive intravenous insulin bolus has been demonstrated to reverse the metabolic state from primary fat utilization to carbohydrate utilization through monitoring of the subject's respiratory quotient.

This study measures whether the reversal of abnormal metabolism in patients with diabetes is correlated with an improvement in their quality of life and associated complication related to their diabetes. The respiratory quotient (RQ) is a measurement of CO2 exhaled and O2 inhaled and is proportionate to the fuel sources being used by the body, primarily the liver over short periods of time. The higher the RQ, the more glucose and less alternative fuel sources are being utilized. Following the RQ change helps determine the effectiveness of physiological intravenous bolus insulin administration in increasing anabolic functions in diabetic individuals. By improving the body's glucose metabolism and thereby causing beneficial effects of anabolic factors, the possibility of serious complications may be decreased. In addition, the use of oral carbohydrate at the same time along with the physiologic intravenous bolus insulin administration stimulates the appropriate gut hormones which augment this effect, a response which cannot be duplicated with intravenous glucose. The purpose of our study is to determine whether the physiologic administration of intravenous bolus insulin along with the augmenting effect of oral carbohydrates will normalize metabolism in diabetic patients and improve their metabolic integrity and quality of life indices.

The RQ is determined by the use of a metabolic cart. Individuals breathe into a mask for 3-5 minutes after a rest period of 20 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQ's higher than 1.05. The RQ can be followed serially to monitor progress aand outcomes and this is done before and after each sixty minute intravenous bolus insulin treatment session, during the 3 successive sessions on a single treatment day. The amount of intravenous insulin and oral glucose given is determined by monitoring the RQ changes during the previous session.Intravenous bolus insulin therapy encourages the glucose metabolism in diabetics to normalize metabolic integrity in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose intravenous insulin boluses similar to those found in non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent glucose levels and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/ VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored every thirty minutes or more frequently as medically necessary to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent intravenous bolus insulin infusion sessions.Patient is evaluated post session and discharged when stable.

Frequent monitoring of RQ and glucose is necessary as these levels change rapidly, depending on the fuel being utilized by the body. Intravenous bolus insulin therapy shifts metabolism from primarily fatty acid metabolism to primarily glucose metabolism. This shift is reflected by the increase in respiratory quotient. However during rest periods the RQ may fall back to lower levels. Therefore RQ's are done at the beginning and at the end of each insulin infusion session of 1 hour in order to appropriately monitor and adjust insulin and carbohydrate loads to reach optimal activation in each session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with significant complications resulting from diabetes
* Ability to swallow without difficulty
* Ability to perform Respiratory Quotient requirements by breathing into a mask for 3 minutes at a time Supervising physician must evaluate and diagnose one of the following medical conditions to be eligible to participate in study
* Hypoglycemia unawareness
* Significant proteinuria (>300 mg/24 hrs) in spite of ACE inhibitors and/or ARB's.
* Diabetic nephropathy
* Progressive, significant diabetic peripheral neuropathy.
* Orthostatic hypotension due to autonomic neuropathy of advanced diabetes.
* Advanced gut neuropathy with gastroparesis or diabetic diarrhea.
* Non-healing diabetic wounds
* Diabetic retinopathy

Exclusion Criteria:

* Lack of intravenous access
* Inability to breathe into a respiratory quotient machine
* Subjects on dialysis
* Presence of severe underlying chronic disease (e.g. coronary artery disease, hepatic disease) which in the opinion of the investigator is likely to preclude the subject from completing the full term of the study
* Inability to stabilize blood pressure at 140/90 or below using ACE inhibitors, Ca channel blockers, Alpha 1 blockers, central Alpha2 agonists or diuretics
* Pregnancy or contemplated pregnancy
* Alcohol abuse, drug addiction or the use of illegal drugs
* Active liver disease
* Active chemotherapy
* Positive HIV
* Subjects with a history of poor compliance to drug or diet or placebo therapy or keeping appointments

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Researchers will assess whether restoring metabolic integrity to diabetic patients improves quality of life and complications associated with diabetes | Patients will have diagnostic testing and complete questionnaires at baseline and every six months thereafter or more frequently if the supervising physician deems medically appropriate throughout the study to monitor and evaluate progress.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cockrell, MD, Principal Investigator — Global Infusion and Aspiration Systems, LLC
Locations (1):
- Global Infusion and Aspiration Systems, LLC, Batesville, Mississippi, United States